CLINICAL TRIAL: NCT05814419
Title: Familial Hyperlipidemia Family Registry
Status: Completed | Type: Observational
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Gary J. Luckasen, MD, Principal Investigator, Poudre Valley Health System
Other Study IDs: 22-1979
Record Dates: First submitted 2023-03-02; First posted 2023-04-14 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Familial Hyperlipidemia
Keywords: Cholesterol; School based; Biometric Screening; Genetic; Healthy Hearts; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
If a child from the Healthy Hearts and Minds education and screening program is found to have a genetic marker for familial hyperlipidemia (FH), immediate family members are offered genetic testing at no charge to identify those at high risk for cardiovascular disorders and those who carry the genetic markers. If identified early, the risk for cardiovascular disease can be greatly modified by early and proper treatment.

The aim of the study is to gauge the impact of large-scale surveillance testing to identify those with the disorder and improve clinical care. This impact is both in disease prevention and in lessening the cost of long-term care from premature cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Primary family member of child from school screening program with documented familial hyperlipidemia (FH) variant

Exclusion Criteria:

* none

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Registry Cohort: If a child from the Healthy Hearts and Minds education and screening program is found to have a genetic marker for familial hyperlipidemia, immediate family members are offered genetic testing at no charge to identify those at high risk for cardiovascular disorders and those who carry the genetic markers. If identified early, the risk for cardiovascular disease can be greatly modified by early and proper treatment. The aim of the study is to gauge the impact of large-scale surveillance testing to identify those with the disorder and improve clinical care. This impact is both in disease prevention and in lessening the cost of long-term care from premature cardiovascular disease.
  Family members of children identified in the Health Hearts screening program were enrolled in this study; Children in the Healthy Hearts screening program were enrolled in NCT05767996
Period: Overall Study
Arm/Group | Observational Registry Cohort
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational Registry Cohort: The aim of the study is to identify children and families that are at risk for cardiovascular disease because of a condition known as familial hyperlipidemia. This condition may increase the risk of cardiac events such as hardening of the arteries anywhere in the body which can result in heart attacks, strokes, and death over ten fold.
  Children have already been assessed in the Healthy Hearts screening program and identified as having elevated cholesterol. A buccal smear will identify whether the familial hyperlipidemia condition exist in your child.
  If the child's test shows that they have the specific gene for familial hyperlipidemia and shows a genetic tendency towards premature heart disease, we would encourage genetic testing for as many blood family members as possible.
  The study plan is to determine whether the Healthy Hearts screening program is a more effective way of identifying students at risk since it is estimated that less than 10% of those individuals with the problem have been identified. If it is effective, then it will be incorporated as part of the standard screening process in the Healthy Hearts program.
Arm/Group | Observational Registry Cohort
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Familial Hypercholesterolemia (FH) Determination for Family Members of School Children With Elevated Cholesterol and Documented FH Variant
Description: Individuals with elevated cholesterol group with familial hypercholesterolemia genotype.
Time Frame: The duration of participation in study is one day.
Population: Individuals with elevated cholesterol group with familial hypercholesterolemia genotype.
  Not enough subjects participating to allow statistical analysis.
Measure: Number; unit: participants
Arm/Group | Observational Registry Cohort
Number analyzed (Participants) | 11
participants
  Positive | 3
  Negative | 8

ADVERSE EVENTS:
Time Frame: There were no adverse events reported during the study from February 17, 2023 (time open to accrual) to May 29, 2025 (time closed to accrual). The only contact with participants was at enrollment so duration was 1 day.
Groups:
- Adverse Events: There were no adverse events reported during the study.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT05814419/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT05814419/ICF_001.pdf